CLINICAL TRIAL: NCT06064175
Title: The Randomized Double-Blind Comparison of Analgesic Efficacy Between Intravenous Forms of Ibuprofen 400 and Ibuprofen 800 mg in Acute Mechanical Low Back Pain in the Emergency Department
Brief Title: "Management of Low Back Pain in the Emergency Department With Different Analgesic Dosages"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Safa Dönmez, M.D., Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Low Back Pain Analgesic
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain, Mechanical; Ibuprofen; Analgesia; Pain Management
MeSH Terms: conditions — Low Back Pain; Agnosia | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen 400 mg-group 1 (Experimental): Patients will receive ibuprofen 400 mg/4 ml via the parenteral route as a rapid 10-minute infusion in 150 ml of saline solution (0.09% NaCl).
  Interventions: Drug: Ibuprofen 400 mg
- Ibuprofen 800 mg-group 2 (Experimental): Patients will receive ibuprofen 800 mg/8 ml via the parenteral route as a rapid 10-minute infusion in 150 ml of saline solution (0.09% NaCl).
  Interventions: Drug: Ibuprofen 800 mg

INTERVENTIONS:
Drug: Ibuprofen 400 mg — Patients will receive ibuprofen 400 mg/4 ml via the parenteral route as a rapid 10-minute infusion in 150 ml of saline solution (0.09% NaCl).
  Arms: Ibuprofen 400 mg-group 1
Drug: Ibuprofen 800 mg — Patients will receive ibuprofen 800 mg/8 ml via the parenteral route as a rapid 10-minute infusion in 150 ml of saline solution (0.09% NaCl).
  Arms: Ibuprofen 800 mg-group 2

SUMMARY:
The Management of Low Back Pain in the Emergency Department Worldwide, low back pain is one of the most prevalent musculoskeletal disorders, and it constitutes one of the primary complaints in emergency departments. A review of the literature reveals studies comparing ibuprofen to various agents (such as paracetamol, nimesulide, acetaminophen), and these studies suggest the use of ibuprofen due to its similar or superior efficacy and its safety profile. However, there is a lack of randomized controlled double-blind comparisons between the commonly recommended single doses of ibuprofen, which are 400 mg and 800 mg. Therefore, the objective of our planned study is to compare the analgesic efficacy of ibuprofen in the forms of 400 mg and 800 mg, which can be administered as a single dose, in the treatment of acute mechanical low back pain, as recommended in all guidelines.

DETAILED DESCRIPTION:
The worldwide prevalence of low back pain makes it one of the most common musculoskeletal disorders, and it ranks among the primary complaints in emergency departments. Literature review reveals studies comparing ibuprofen to various agents (such as paracetamol, nimesulide, acetaminophen), and these studies suggest the use of ibuprofen due to its similar or superior efficacy and its safety profile. However, there is a lack of randomized controlled double-blind comparisons between the commonly recommended single doses of ibuprofen, which are 400 mg and 800 mg. Therefore, the objective of our planned study is to compare the analgesic efficacy of ibuprofen in the forms of 400 mg and 800 mg, which can be administered as a single dose, in the treatment of acute mechanical low back pain, as recommended in all guidelines.

The expected benefit of the research is to determine whether the analgesic effectiveness of ibuprofen 400 mg is equivalent to that of 800 mg, thereby potentially reducing the unnecessary use of higher doses of NSAIDs. Alternatively, if the 800 mg parenteral form proves to be more effective, it may suggest recommending the standard single-dose use of 800 mg for analgesia in acute mechanical low back pain.

The research is designed as a prospective, randomized-double-blind, single-center study.

The study is divided into two arms, labeled as Arm 1 and Arm 2. Randomization will be conducted by the principal investigator. For patients who agree to participate in the study, pre-assigned medications will be administered using a computer program. The relevant medications will be numbered and placed in envelopes within this computer program, which will then be labeled as Treatment 1 and Treatment 2. The randomly selected medication (Treatment 1 or Treatment 2) will be administered by a nurse, and the administering nurse will subsequently be separated from the patient's treatment and follow-up.

Upon the arrival of a patient who meets the inclusion criteria, the informed consent form will be obtained. The patient will be assigned to the research arm according to the randomization scheme. Research arms are divided into Arm 1 and Arm 2. In both arms, ibuprofen solutions of 400 mg/4 ml and 800 mg/8 ml will be prepared and administered as rapid infusions over 10 minutes in 150 ml of saline solution (0.09% NaCl).

After the patient arrives, the attending physician will inform the nurse that a patient is being enrolled in the study. The nurse will prepare the injector as specified in the order. The patient will be asked to mark their pain level on a 10-point NRS before injection. They will be asked to mark their pain level again at 15, 30, 60, and 120 minutes. If there is no relief in pain level by the 30th minute or if the pain level does not decrease to the desired level (NRS>3) at 60 or 120 minutes, rescue medication will be administered.

The rescue medication protocol will involve tramadol citrate 100 mg. It will be administered as an intravenous infusion in 500 cc of normal saline over 20-30 minutes to minimize possible side effects and ensure controlled delivery.

If the patient wishes to withdraw from the study during this follow-up period or if any complications arise, they will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above but under 65 years old.
* Patients willing to participate in the study.
* Patients with acute pain lasting less than two weeks.
* Non-traumatic pain.
* Patients without radicular back pain.
* Patients scoring more than 5 points on the 24-item validated Roland Morris Disability Questionnaire (RMDQ).
* Patients marking more than 4 on the Numeric Pain Rating Scale (NRS).
* Patients deemed appropriate for the study by an emergency medicine specialist based on history and physical examination.
* Patients in whom other differential diagnoses are not primarily considered.

Exclusion Criteria:

* - Patients aged below 18 and above 65.
* Patients who decline to participate in the study.
* Patients with vital signs outside normal limits.
* Patients with a history of adverse reactions to ibuprofen.
* Patients unable to determine their pain intensity on the NRS.
* Pregnant individuals.
* Individuals with a history of heart disease and hypertension.
* Individuals with advanced systemic diseases.
* Patients with malignancies.
* Patients with chronic liver disease.
* Individuals using neuro-psychiatric drugs with sedative and analgesic effects.
* Individuals with a history of psychological and neurological diseases.
* Patients who used analgesics within 6 hours before examination.
* Patients with pain lasting more than two weeks.
* Traumatic cases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
NRS | 15., 30., 60. and 120. minutes
  Numeric Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: SAFA DÖNMEZ, M.D., Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not have a data sharing plan for this study; however, the data set will be shared upon publication with the journal that has been submitted to.

REFERENCES:
- [Background] Oliveira IS, Vanin AA, Pena Costa LO, Medeiros FC, Ananias Oshima RK, Inacio AA, Matos da Cunha TA, Palomo AS, Fukuda TY, de Freitas DG, Benvenuto F, Menezes Costa LDC. Profile of Patients With Acute Low Back Pain Who Sought Emergency Departments: A Cross-sectional Study. Spine (Phila Pa 1976). 2020 Mar 1;45(5):E296-E303. doi: 10.1097/BRS.0000000000003253. PMID 32045404
- [Background] Ostojic P, Radunovic G, Lazovic M, Tomanovic-Vujadinovic S. Ibuprofen plus paracetamol versus ibuprofen in acute low back pain: a randomized open label multicenter clinical study. Acta Reumatol Port. 2017 Jan-Mar;42(1):18-25. PMID 27978532
- [Background] Friedman BW, Irizarry E, Chertoff A, Feliciano C, Solorzano C, Zias E, Gallagher EJ. Ibuprofen Plus Acetaminophen Versus Ibuprofen Alone for Acute Low Back Pain: An Emergency Department-based Randomized Study. Acad Emerg Med. 2020 Mar;27(3):229-235. doi: 10.1111/acem.13898. Epub 2020 Jan 7. PMID 31811673
- [Background] Pohjolainen T, Jekunen A, Autio L, Vuorela H. Treatment of acute low back pain with the COX-2-selective anti-inflammatory drug nimesulide: results of a randomized, double-blind comparative trial versus ibuprofen. Spine (Phila Pa 1976). 2000 Jun 15;25(12):1579-85. doi: 10.1097/00007632-200006150-00019. PMID 10851109
- [Background] Tuzun F, Unalan H, Oner N, Ozguzel H, Kirazli Y, Icagasioglu A, Kuran B, Tuzun S, Basar G. Multicenter, randomized, double-blinded, placebo-controlled trial of thiocolchicoside in acute low back pain. Joint Bone Spine. 2003 Sep;70(5):356-61. doi: 10.1016/s1297-319x(03)00075-7. PMID 14563464